# Statistical Analysis Plan

Obstructive Sleep Apnea in WTC responders: Role of nasal Pathology

NCT01753999

January 03, 2020

### **Primary Outcome Measure: Measure Title Adherence to CPAP**

Measure Description: The use (number of hours per night) will be compared between standard CPAP and CPAP flex.

#### Statistical method:

Generalized estimating equations (GEE) models, with mean hours per night as the dependent variable, will be used to compare the device use of standard CPAP and CPAP flex.

## **Secondary Outcome Measure: Measure Title CPAP Efficacy**

Measure Description: Efficacy will be evaluated by measuring the apnea and hypopnea index (AHI) during treatment. The efficacy of standard CPAP and CPAP flex will be compared.

#### Statistical method:

Generalized estimating equations (GEE) models, with AHI as the dependent variable, will be used to compare the efficacy between standard CPAP and CPAP flex.